CLINICAL TRIAL: NCT05721014
Title: Effects of OsteoStrong vs. Individually Adapted and Combined Training on Bone Health Amongst Older Women With High Fracture Risk: A Randomised Controlled Trial
Brief Title: Effects of OsteoStrong vs. Individually Adapted and Combined Training on Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); The Swedish School of Sport and Health Sciences (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Helena Salminen, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04359 Osteostrong
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis; Osteopenia; Bone Density, Low; Bone Loss
Keywords: osteoporosis; osteopenia; bone mineral density; bone density; physical activity; strength training; isometric training
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OsteoStrong (Experimental): Training following the OsteoStrong-method.
  Interventions: Other: OsteoStrong
- Individually Adapted and Combined Physical Training (Active Comparator): Training based on current recommendations on exercise for people with osteoporosis.
  Interventions: Other: Individually Adapted and Combined Physical Training

INTERVENTIONS:
Other: OsteoStrong — This training method is an isometric high-impact loading in four different training machines (Spectrum) and balance training on a vibration plate. The four machines are "chest press", "leg press", "pull-down" and "deadlift". The participants press and/or pull isometrically for around 10-15 seconds 1-3 times on every machine.
  The training session takes around 20 minutes and is performed individually by the participants with the help of a training instructor.
  Arms: OsteoStrong
Other: Individually Adapted and Combined Physical Training — This training method is based on the current recommendations on physical activity for people with osteoporosis.
  The training is divided into two training sessions:
  Circuit training with ten stations with different exercises for the whole body (strength, balance, endurance, weight-bearing). The participants spend 40 seconds on each station. This is repeated during 40 minutes. The training session starts with a joint warm-up and ends with a cool-down.
  Strength training with machines for the whole body with the intensity of up to 70-80 % of one repetition max (1RM). The training session starts with a joint warm-up and and a voluntary individual cool-down.
  The training session takes around 60 minutes and is performed in a group with the help of a training instructor. The participants also have the option to do a home based exercise programme that they could do in a few cases when they were unable to attend the physical group training.
  Arms: Individually Adapted and Combined Physical Training

SUMMARY:
The aim of this clinical trial is to investigate the effect of the OsteoStrong training method and the Individually Adapted and Combined Training on the bone health of older women with high fracture risk. Additionally, the aim is also to explore the participants' experiences of each training method.

Participants will be randomised to either treatment arm A (OsteoStrong) or treatment arm B (Individually Adapted and Combined Training). Participants in both groups will train for nine months. Treatment arm A will train individually once a week and treatment arm B will train in a group twice a week. Both groups will have a training instructor who will supervise and give training instructions.

Researchers will compare the groups to see the effects of the training methods on the participants' bone health among other outcome measures. The participants will be tested at baseline and post-intervention (9 months later).

ELIGIBILITY:
Inclusion Criteria:

* Woman, 65-79 years old.
* Vaccinated against Covid-19.
* Be able to participate in nine months of training.
* Untreated with Osteoporosis-medications, or have an ongoing treatment since at least one year back.

Exclusion Criteria:

* Ongoing treatment with Osteoporosis-medications with an onset within a year, or a previous treatment which was terminated within the last five years.
* Ongoing treatment with Osteoporosis-medications that has been delayed for more than eight months for Denosumab, or more than 18 months for bisphosphonates.
* Vertebral fracture, that have been diagnosed within three months.
* Vertebral fracture or hip fracture, that have not previously been treated with Osteoporosis-medications or been assessed by a physician.
* Bilateral hip replacements.
* Symptomatic disc herniation, inguinal herniation or umbilical herniation.
* Untreated hypertension.
* Other diseases that can affect the results and participation in the study: malignant diseases, muscle dystrophy, secondary osteoporosis, or other conditions that would hinder study participation.
* Ongoing treatment with oral cortisone pills (≥ 5 mg Prednisolone).
* Conditions that hinders the conduction of impact microindentation with OsteoProbe: large edema, skin infection, allergy towards local anaesthetics.
* Ongoing or previous training (within the last year) at OsteoStrong.

Ages: 65 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Bone Material Strength Index (BMSI) | Change from baseline at 9 months
  Bone Material Strength Index measured with impact microindentation using OsteoProbe

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) | Change from baseline at 9 months
  Bone Mineral Density and T-score measured with Dual-Energy X-ray Absorptiometry (DXA)
Procollagen Type 1 N-terminal propeptide (S-PINP) | Change from baseline at 3 and 9 months
  Bone biomarker
Serum C-telopeptide cross-link type 1 collagen (S-CTX) | Change from baseline at 3 and 9 months
  Bone biomarker
Sclerostin | Change from baseline at 3 and 9 months
  Bone biomarker
Bone alkaline phosphatase (S-BALP) | Change from baseline at 3 and 9 months
  Bone biomarker
Self-rated health questionnaire (SF-36) | Change from baseline at 9 months
  A questionnaire with multiple choice questions about general health
Falls Efficacy Scale (FES) | Change from baseline at 9 months
  A questionnaire about self-efficacy and fear of falling, 1-10, where 0 equals "not sure at all" and 10 equals "completely sure". Higher scores equals better outcome.
Socialstyrelsens questionnaire for lifestyle habits | Change from baseline at 9 months
  A questionnaire with multiple choice questions about falls and fractures, physical activity, sitting, alcohol and smoking
Numerical Rating Scale (NRS) | Change from baseline at 3 and 9 months
  A pain rating scale from 0-10, where 0 equals "no pain" and 10 equals "maximum/worst possible pain imaginable". Higher scores equals worse outcome.
Back extension strength | Change from baseline at 9 months
  Measuring back extension strength with Digimax
Grip strength | Change from baseline at 9 months
  Measuring grip strength with hand dynamometer (JAMAR)
Chair stand test | Change from baseline at 9 months
  5 seconds, 30 seconds and time for making 50 chair stands
Back extension endurance | Change from baseline at 9 months
  Measuring back extension endurance with Sörensen's test
Static sit-up | Change from baseline at 9 months
  Sitting with the upper body in 45 degrees
Lung capacity | Change from baseline at 9 months
  Lung capacity measured with dynamic spirometry (Welch Allyn)
One leg standing (eyes open) | Change from baseline at 9 months
  Balance test
One leg standing (eyes closed) | Change from baseline at 9 months
  Balance test
Two leg standing on a straight line (eyes open) | Change from baseline at 9 months
  Balance test
Two leg standing on a straight line (eyes closed) | Change from baseline at 9 months
  Balance test
Walking forward on a straight line | Change from baseline at 9 months
  Balance test
Walking backwards between to lines | Change from baseline at 9 months
  Balance test
BtrackS | Change from baseline at 9 months
  Balance test, measuring body sway, standing on a platform with both legs together, arms crossed and eyes closed.
Accelerometry | Change from baseline at 9 months
  Accelerometers worn around the waist to measure physical activity levels for up to nine days.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Salminen, Ass. prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet - Department of Neurobiology, Care Sciences and Society: Division of Family medicine and Primary care, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The website for the study. — https://ki.se/nvs/den-benstarka-studien-kan-vi-med-traning-starka-vart-skelett